CLINICAL TRIAL: NCT02277444
Title: A Multicenter, Open-Label Trial of Intravenous Golimumab, a Human Anti-TNFα Antibody, in Pediatric Subjects With Active Polyarticular Course Juvenile Idiopathic Arthritis Despite Methotrexate Therapy
Brief Title: A Study to Evaluate the Pharmacokinetics, Efficacy and Safety of Intravenous Golimumab in Pediatric Participants With Active Polyarticular Course Juvenile Idiopathic Arthritis Despite Methotrexate Therapy
Acronym: GO-VIVA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR105178; CNTO148JIA3003 (Other: Janssen Research & Development, LLC); 2015-004804-47 (EudraCT Number)
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Arthritis, Juvenile
Keywords: Methotrexate; Anti-TNFα Antibody; Golimumab; Pediatric Participants
MeSH Terms: conditions — Arthritis, Juvenile | interventions — golimumab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Golimumab + Methotrexate (Experimental): Participants will receive 80 milligram per meter square (mg/m^2) as an intravenous (IV) infusion at Weeks 0, 4, and every 8 weeks thereafter up to Week 244, along with commercial methotrexate (MTX) weekly through Week 28 at the same Body Surface Area (BSA)-based dosage (10 to 30 mg/m^2 per week for participants with BSA less than [<] 1.67 meter square (m^2), or minimum of 15 mg/week for participants with BSA greater than or equal to [>=] 1.67 m^2) as at the time of study entry. At Week 252, participants who meet the criteria for the optional Extended Treatment Period (ETP) may continue treatment with golimumab 80 mg/m^2 every 8 weeks after completion of the Week 252 assessments.
  Interventions: Drug: Golimumab; Drug: Methotrexate

INTERVENTIONS:
Drug: Golimumab — Golimumab 80 mg/m^2 IV infusion at Weeks 0, 4, and every 8 weeks through Week 244. At Week 252, participants who meet the criteria for the optional Extended Treatment Period (ETP) may continue treatment with golimumab 80 mg/m^2 every 8 weeks after completion of the Week 252 assessments.
  Other Names: Simponi Aria
Drug: Methotrexate — Methotrexate BSA-based dose (10 to 30 mg/m^2 per week for participants with BSA <1.67 m^2, or minimum of 15 mg/week for participants with BSA >=1.67 m^2) weekly at least through Week 28.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (the study of the way a drug enters and leaves the blood and tissues over time) of golimumab administered intravenously (IV) to pediatric participants with polyarticular (affects 5 or more joints) juvenile (an onset before age 16) idiopathic (of unknown cause) arthritis (joint pain) (pJIA) manifested by greater than or equal to (>=) 5 joints with active arthritis despite methotrexate (MTX) therapy for >= 2 months.

DETAILED DESCRIPTION:
This is a single arm, Open-label (all people know the identity of the intervention), multi-center (when more than one hospital or medical school team work on a medical research study) study to determine the pharmacokinetics (the study of the way a drug enters and leaves the blood and tissues over time), efficacy (effectiveness) and safety of intravenous golimumab in participants with pJIA despite current treatment with methotrexate (MTX). The study will consist of 3 parts: Screening Phase (6 weeks); an Open-label Treatment Phase (consists of golimumab and MTX treatment for 52 weeks, wherein after Week 28, MTX dose change is allowed); Long-term Extension Phase (after Week 52 through Week 252) and Extended Treatment Period (after week 252). The maximal study duration for a participant will not exceed 832 weeks. All the eligible participants will be administered golimumab IV infusion and commercial MTX. Blood samples will be collected for evaluation of pharmacokinetics of study treatment. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis must be made per Juvenile Idiopathic Arthritis (JIA) International League of Associations for Rheumatology (ILAR) diagnostic criteria and the onset of disease must have been before the participant's 16th birthday
* Failure or inadequate response to at least a 2 month course of methotrexate (MTX) before screening
* Participants must have greater than or equal to (>=) 5 joints with active arthritis at screening and at Week 0 as defined by American College of Rheumatology (ACR) criteria (that is, a joint with either swelling, or in the absence of swelling, limited range of motion associated with pain on motion or tenderness)
* Participants must have a screening C-reactive protein (CRP) of >=0.1 milligram (mg)/deciliter (dL) with the exception of approximately 30 percent (%) of the study population
* Participants must have active polyarticular juvenile idiopathic arthritis (pJIA) despite current use of oral, intramuscular, or subcutaneous MTX for >=2 months before screening. For participants with body surface area (BSA) less than (<)1.67 meter square (m^2), the MTX dose must be between 10 to 30 milligram per meter square (mg/m^2) per week and stable for >=4 weeks before screening. For participants with BSA >=1.67 m^2, the MTX dose must be a minimum of 15 mg/week and must be stable for >=4 weeks before screening. In situations where there is documented intolerance of doses greater than (>)10 mg/m^2 weekly (for participants with BSA <1.67 m^2) or >=15 mg/week (for participants with BSA >=1.67 m^2); or where documented country or site regulations prohibit use of >=15 mg of MTX per week in participants with BSA >=1.67 m^2, participants may be entered into the trial on a lower dose of MTX

Exclusion Criteria:

* Participant has initiated disease-modifying antirheumatic drugs (DMARDs) and/or immunosuppressive therapy within 4 weeks prior to first study agent administration
* Participant has been treated with intra-articular, intramuscular or intravenous corticosteroids (including intramuscular corticotropin) during the 4 weeks before first study agent administration
* Participant has been treated with any therapeutic agent targeted at reducing Interleukin (IL)-12 or IL 23, including but not limited to ustekinumab and ABT-874, within 3 months before first study agent administration
* Participant has been treated with natalizumab, efalizumab, or therapeutic agents that deplete B or T cells (eg, rituximab, alemtuzumab, or visilizumab) during the 12 months before first study agent administration, or have evidence at screening of persistent depletion of the targeted lymphocyte after receiving any of these agents
* Participant has been treated with alefacept within 3 months before first study agent administration
* If a participant has been previously treated with an anti-tumor necrosis factor alpha (TNF alpha) agent, the reason for discontinuation of the anti-TNF alpha agent cannot have been a severe or serious adverse event consistent with the class of anti-TNF alpha agents

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2014-12-22 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2024-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (38):
- United States (14):
  - San Diego, California
  - Chicago, Illinois
  - Boston, Massachusetts
  - Hackensack, New Jersey
  - New Hyde Park, New York
  - Durham, North Carolina
  - Hickory, North Carolina
  - Avon, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - Salt Lake City, Utah
- Argentina (3):
  - Buenos Aires
  - Rosario
  - San Miguel de Tucumán
- Brazil (5):
  - Botucatu
  - Campinas
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
- Canada (3):
  - Calgary, Alberta
  - Toronto, Ontario
  - Montreal, Quebec
- Región Metropolitana de Santia, Chile
- Israel (3):
  - Haifa
  - Kfar Saba
  - Petah Tikva
- Mexico (3):
  - Chihuahua City
  - Guadalajara
  - Mexico City
- Russia (5):
  - Mosco2
  - Saint Petersburg
  - Saratov
  - Tolyatti
  - Ufa
- Cape Town, South Africa

REFERENCES:
- [Derived] Leu JH, Shiff NJ, Clark M, Bensley K, Lomax KG, Berezny K, Nelson RM, Zhou H, Xu Z. Intravenous Golimumab in Patients with Polyarticular Juvenile Idiopathic Arthritis and Juvenile Psoriatic Arthritis and Subcutaneous Ustekinumab in Patients with Juvenile Psoriatic Arthritis: Extrapolation of Data from Studies in Adults and Adjacent Pediatric Populations. Paediatr Drugs. 2022 Nov;24(6):699-714. doi: 10.1007/s40272-022-00533-y. Epub 2022 Sep 28. PMID 36171515
- [Derived] Ruperto N, Brunner HI, Pacheco-Tena C, Louw I, Vega-Cornejo G, Spindler AJ, Kingsbury DJ, Schmeling H, Borzutzky A, Cuttica R, Inman CJ, Malievskiy V, Scott C, Keltsev V, Terreri MT, Viola DO, Xavier RM, Fernandes TAP, Velazquez MDRM, Henrickson M, Clark MB, Bensley KA, Li X, Lo KH, Leu JH, Hsu CH, Hsia EC, Xu Z, Martini A, Lovell DJ; Pediatric Rheumatology Collaborative Study Group (PRCSG) and the Paediatric Rheumatology International Trials Organisation (PRINTO). Open-label phase 3 study of intravenous golimumab in patients with polyarticular juvenile idiopathic arthritis. Rheumatology (Oxford). 2021 Oct 2;60(10):4495-4507. doi: 10.1093/rheumatology/keab021. PMID 33493312

RESULTS

PARTICIPANT FLOW:
Groups:
- Golimumab: Participants received 80 milligrams per meter square (mg/m^2) golimumab as an intravenous (IV) infusion at Weeks 0, 4, and then every 8 weeks (q8w) till Week 52. Participants also received commercial methotrexate (MTX) weekly through Week 28 at the same body surface area (BSA)-based dosage (10 to 30 mg/m^2 per week for participants with BSA less than [<] 1.67 meter square [m^2], or minimum of 15 mg/week for participants with BSA greater than or equal to [>=] 1.67 m^2) as at time of study entry. After Week 28, changes in MTX administration were permitted. Participants who completed Week 52 had the option to enter into the long-term extension (LTE) phase. Participants who opted not to enter the LTE completed an additional 8-week safety follow-up visit following the last administration of the study agent. Participants who entered LTE continued to receive 80 mg/m^2 IV golimumab q8w through Week 244. All participants who completed Week 244 were followed for safety through Week 252. Participants who met the inclusion criteria entered the extended treatment period (ETP) and continued to receive 80 mg/m^2 IV golimumab q8w from Week 252 to Week 420.
Period: Treatment Period (Week 0-52)
Arm/Group | Golimumab
Started | 130
Treated | 127
Completed | 112
Not Completed | 18
Not completed — Adverse Event | 11
Not completed — Withdrawal by Subject | 3
Not completed — Other | 1
Not completed — Enrolled and not Treated | 3
Period: LTE Period (Week 52 to Week 252)
Arm/Group | Golimumab
Started | 112
Completed | 69
Not Completed | 43
Not completed — Other | 43
Period: ETP Period (Week 252 to Week 420)
Arm/Group | Golimumab
Started (Participants who completed the study through Week 252, for whom the drug was found to be beneficial but was not commercially available for polyarticular juvenile idiopathic arthritis, were enrolled in the ETP at Week 252.) | 32
Completed | 18
Not Completed | 14
Not completed — Adverse Event | 1
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 2
Not completed — Other | 8

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least 1 dose of study agent.
Arm/Group | Golimumab
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.6 (3.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 1
  Black or African American | 5
  More than one race | 4
  Other | 28
  White | 85
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 18
  BRAZIL | 16
  CANADA | 7
  CHILE | 7
  ISRAEL | 2
  MEXICO | 25
  RUSSIAN FEDERATION | 14
  SOUTH AFRICA | 15
  UNITED STATES | 23

OUTCOME MEASURES:

1. Primary Outcome: Serum Trough Concentration (C-trough) of Golimumab
Description: Serum golimumab trough concentration at Week 28 was reported.
Time Frame: Week 28
Population: The pharmacokinetic (PK) analysis set included all treated participants (who received at least 1 infusion) who have sufficient PK samples for analysis. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Golimumab
Number analyzed (Participants) | 87
micrograms per milliliter (mcg/mL) | 0.50 (0.427)

2. Primary Outcome: Bayesian Area Under Curve at Steady State (AUCss) Over an 8-week Dosing Interval at Week 28
Description: AUCss was defined as area under the plasma concentration-time curve at steady-state (based on steady-state assessment of trough concentrations or via modeling).
Time Frame: Week 28
Population: The PK analysis set included all treated participants (who received at least 1 infusion) who have sufficient PK samples for analysis.
Measure: Median (Full Range); unit: micrograms*day/milliliter (mcg*day/mL)
Arm/Group | Golimumab
Number analyzed (Participants) | 127
micrograms*day/milliliter (mcg*day/mL) | 399 [387 to 424]

3. Secondary Outcome: Serum Trough Concentration (C-trough) at Week 52
Description: Serum golimumab trough concentration at Week 52 was reported.
Time Frame: Week 52
Population: The PK analysis set included all treated participants (who received at least 1 infusion) who have sufficient PK samples for analysis. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Golimumab
Number analyzed (Participants) | 95
mcg/mL | 0.52 (0.475)

4. Secondary Outcome: Baysesian Area Under Curve at Steady State (AUCss) at Week 52
Description: as for outcome 2
Time Frame: Week 52
Population: as for outcome 2
Measure: Median (Full Range); unit: mcg*day/mL
Arm/Group | Golimumab
Number analyzed (Participants) | 127
mcg*day/mL | 421 [402 to 446]

ADVERSE EVENTS:
Time Frame: Treatment Period Arm: All cause mortality (From screening [-6 weeks] up to Week 52), Serious and Other AEs (Week 0 up to Week 52); LTE Period Arm: Week 52 up to Week 252; ETP Arm: Week 252 up to Week 420
Description: All Cause mortality reported for all randomized participants. Serious and other AEs: The full analysis set includes all enrolled participants who received at least 1 infusion.
Groups:
- Treatment Period (Week 0 to 52): Golimumab 80 mg/m^2 IV q8w: Participants received 80 milligrams per meter square (mg/m^2) golimumab as an intravenous (IV) infusion at Weeks 0, 4, and then every 8 weeks (q8w) till Week 52. Participants also received commercial methotrexate (MTX) weekly through Week 28 at the same body surface area (BSA)-based dosage (10 to 30 mg/m^2 per week for participants with BSA less than [<] 1.67 meter square [m^2], or minimum of 15 mg/week for participants with BSA greater than or equal to [>=] 1.67 m^2) as at time of study entry. After Week 28, changes in MTX administration were permitted. Participants who completed Week 52 had the option to enter into the long-term extension (LTE) phase.
- LTE Period (Week 52 to 252): Golimumab 80 mg/m^2 IV q8w: Participants who completed Week 52 and entered into the LTE phase, continued to receive 80 mg/m^2 intravenous golimumab every 8 weeks through Week 244. Those who chose not to enter LTE completed an additional 8-week safety follow-up visit after their final administration of the study agent. All participants who completed Week 244 were monitored for safety through Week 252.
- ETP (Week 252 to 420): Golimumab 80 mg/m^2 IV q8w: Participants who met the inclusion criteria entered the ETP and continued receiving 80 mg/m^2 intravenous golimumab every 8 weeks from Week 252 to Week 420.
Arm/Group | Treatment Period (Week 0 to 52): Golimumab 80 mg/m^2 IV q8w | LTE Period (Week 52 to 252): Golimumab 80 mg/m^2 IV q8w | ETP (Week 252 to 420): Golimumab 80 mg/m^2 IV q8w
All-Cause Mortality (participants affected / at risk) | 1/127 | 1/127 | 0/32
Serious Adverse Events (participants affected / at risk) | 9/127 | 18/127 | 3/32
Other Adverse Events (participants affected / at risk) | 74/127 | 57/127 | 8/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period (Week 0 to 52): Golimumab 80 mg/m^2 IV q8w (N=127) | LTE Period (Week 52 to 252): Golimumab 80 mg/m^2 IV q8w (N=127) | ETP (Week 252 to 420): Golimumab 80 mg/m^2 IV q8w (N=32)
Myopericarditis (Cardiac disorders) | 0 | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Retinal Detachment (Eye disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Crohn's Disease (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Calcinosis (General disorders) | 0 | 1 | 1
Drug Intolerance (General disorders) | 0 | 1 | 0
Ocular Implant Exposure (General disorders) | 0 | 0 | 1
Temperature Regulation Disorder (General disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1 | 0
Disseminated Tuberculosis (Infections and infestations) | 0 | 1 | 0
Escherichia Infection (Infections and infestations) | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0
Herpes Zoster Disseminated (Infections and infestations) | 1 | 0 | 0
Infective Exacerbation of Bronchiectasis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Pneumonia Streptococcal (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Septic Shock (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Varicella (Infections and infestations) | 1 | 1 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cutaneous T-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Generalised Anxiety Disorder (Psychiatric disorders) | 0 | 1 | 0
Major Depression (Psychiatric disorders) | 0 | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cyanosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period (Week 0 to 52): Golimumab 80 mg/m^2 IV q8w (N=127) | LTE Period (Week 52 to 252): Golimumab 80 mg/m^2 IV q8w (N=127) | ETP (Week 252 to 420): Golimumab 80 mg/m^2 IV q8w (N=32)
Abdominal Pain (Gastrointestinal disorders) | 8 | 2 | 0
Nausea (Gastrointestinal disorders) | 11 | 7 | 0
Vomiting (Gastrointestinal disorders) | 10 | 5 | 0
Gastroenteritis (Infections and infestations) | 6 | 12 | 1
Nasopharyngitis (Infections and infestations) | 22 | 16 | 2
Pharyngitis (Infections and infestations) | 4 | 8 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 28 | 19 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 12 | 0
Alanine Aminotransferase Increased (Investigations) | 7 | 1 | 0
Arthritis (Nervous system disorders) | 4 | 7 | 3
Juvenile Idiopathic Arthritis (Musculoskeletal and connective tissue disorders) | 14 | 18 | 2
Headache (Nervous system disorders) | 14 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT02277444/Prot_002.pdf
  • Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT02277444/SAP_003.pdf